CLINICAL TRIAL: NCT03099954
Title: Withings Pulse Wave Velocity and Blood Pressure Study
Status: Completed | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Collaborators: Withings (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB-16-6856
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2017-06

CONDITIONS: Elevated Blood Pressure; Hypertension; Mental Stress; Sleep Disorders
MeSH Terms: conditions — Hypertension; Stress, Psychological; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Measure pulse wave velocity stability in relation to time of day, day of the week, physical activity, sleep quality, stress levels and blood pressure.

DETAILED DESCRIPTION:
The study population will be an estimated 300 healthy adult subjects from the United States. This population will be approximately 150 men and 150 women. In order to obtain a relatively diverse age range of users (with varying levels of arterial stiffness), we hope to enroll participants across three age ranges entered in the Withings application by the user: 18-40 years, 41-60 years, and > 60 years. These spots will be filled by those that satisfy the inclusion/exclusion criteria on a first come, first served basis.

ELIGIBILITY:
Inclusion Criteria:

* User of a (1) Withings blood pressure cuff (2) Withings activity tracker and (3) Withings Body Cardio scale
* User has measured their blood pressure at least once per week for the majority of weeks over the last three months.

Exclusion Criteria:

* Aortic artery disease
* Peripheral vascular disease
* Atrial fibrillation
* Weight > 396 lbs.
* Pregnant women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will be an estimated 300 healthy adult subjects from the United States. This population will be approximately 150 men and 150 women
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Measure pulse wave velocity (PWV) stability in relation to time of day, day of the week, physical activity, sleep quality, stress levels and blood pressure. | Subjects will be expected to participate for a total of 16 weeks.
  The study population will be an estimated 300 healthy adult subjects from the United States who own a Withings blood pressure cuff, Withings activity tracker, and Withings Body Cardio scale and have measured their blood pressure at least once per week for the majority of weeks over the last three months.

CONTACTS AND LOCATIONS:
Overall Officials: Brian D Modena, MD, Principal Investigator — Scripps Translational Science Institute
Locations (1):
- Scripps Translational Science Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided